CLINICAL TRIAL: NCT02857335
Title: Neurocognitive Outcome in Children Who Suffered From Idiopathic Increased Intracranial Hypertension (IIH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HYMC-0100-15
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Prospective Study , Questionaires
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study group (Other): patients with benign intracranial hypertension ages 8-16 years
  Interventions: Behavioral: neurocognitive tests

INTERVENTIONS:
Behavioral: neurocognitive tests — Subjects will undergoe a battery of neurocognitive testing which will test memory, flexible thought process, problem, attention span

SUMMARY:
15 patients, Ages 8-17 who were diagnosed in the recent years with Idiopathic increased intracarnial hypertension (IIH) went through a battery of neurocognitive tests to establish whether there was any affect of the disease on their cognitive function

ELIGIBILITY:
Inclusion Criteria:

* children who suffered from IIH based on history, physical examination, ophtalmological exam, LP results, Brain imagining

Exclusion Criteria:

* co morbidities

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
neurocognitive outcomes | once
  The computerized battery of tests used in this study (testing time: 30 minutes) sampled non-verbal memory, executive function, visual spatial processing, attention, motor skills, problem solving, and information processing speed. Outcome parameters for tests or test levels included accuracy, reaction time (RT), standard deviation (SD) of RT, and a composite score ([accuracy/RT] · 100). Normalized subsets of outcome parameters were averaged to produce 7 summary scores. The outcome parameters contributing to each index score were included. The Global Cognitive Score (GCS) was computed as the average of the index scores.

SECONDARY OUTCOMES:
Non-Verbal Memory | once
  Eight pictures of simple geometric objects were presented, followed by a recognition test, in which 4 versions of each object were presented, each oriented in a different direction
Go-No Go Test | once
  A series of large colored stimuli were presented at pseudorandom intervals. Participants were instructed to respond as quickly as possible by pressing a mouse button if the color of the stimulus was any color except red, for which no response was made
Stroop Interference | once
  Participants were presented with a pair of large colored squares, one on the left and the other on the right side of the screen. In each phase, the participants were instructed to choose as quickly as possible which of the 2 squares was a particular color.
Visual Spatial Processing | once
  Computer-generated scenes containing a red pillar were presented. Participants were instructed to imagine viewing the scene from the vantage point of the red pillar. Four alternative views of the scene were shown as choices
Staged Information Processing Speed | once
  comprises 3 levels of information processing load: single digits, 2-digit arithmetic problems.For each of the 3 levels, stimuli were presented at 3 different fixed rates, incrementally increasing as testing continues.
cognitive domains | once
  Participants had to "catch" a rectangular white object falling vertically from the top of the screen before it reached the bottom of the screen. Pressing on the mouse button moved a rectangular green "paddle" horizontally so that it could be positioned directly in the path of the falling object. The test required hand-eye coordination, scanning, and rapid responses
Problem Solving | once
  Pictorial puzzles of gradually increasing difficulty were presented. Each puzzle consisted of a 2 · 2 array containing 3 black and white line drawings and a missing element. Participants had to choose the best fit for the fourth (missing) element of the puzzle from among 6 possible alternatives.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] D'Amico D, Curone M, Erbetta A, Farago' G, Bianchi-Marzoli S, Ciasca P, Bussone G, Chiapparini L. Intracranial idiopathic hypertension: 1-year follow-up study. Neurol Sci. 2014 May;35 Suppl 1:177-9. doi: 10.1007/s10072-014-1765-x. PMID 24867861
- [Background] Wall M. Idiopathic intracranial hypertension. Neurol Clin. 2010 Aug;28(3):593-617. doi: 10.1016/j.ncl.2010.03.003. PMID 20637991
- [Background] Dave SB, Subramanian PS. Pseudotumor cerebri: an update on treatment options. Indian J Ophthalmol. 2014 Oct;62(10):996-8. doi: 10.4103/0301-4738.145991. PMID 25449933
- [Background] Afonso CL, Talans A, Monteiro ML. Factors affecting visual loss and visual recovery in patients with pseudotumor cerebri syndrome. Arq Bras Oftalmol. 2015 May-Jun;78(3):175-9. doi: 10.5935/0004-2749.20150045. PMID 26222108
- [Background] Zur D, Naftaliev E, Kesler A. Evidence of multidomain mild cognitive impairment in idiopathic intracranial hypertension. J Neuroophthalmol. 2015 Mar;35(1):26-30. doi: 10.1097/WNO.0000000000000199. PMID 25383589
- [Background] Kharkar S, Hernandez R, Batra S, Metellus P, Hillis A, Williams MA, Rigamonti D. Cognitive impairment in patients with Pseudotumor Cerebri Syndrome. Behav Neurol. 2011;24(2):143-8. doi: 10.3233/BEN-2011-0325. PMID 21606575
- [Background] Soiberman U, Stolovitch C, Balcer LJ, Regenbogen M, Constantini S, Kesler A. Idiopathic intracranial hypertension in children: visual outcome and risk of recurrence. Childs Nerv Syst. 2011 Nov;27(11):1913-8. doi: 10.1007/s00381-011-1470-5. Epub 2011 May 3. PMID 21538129
- See also: Related Info — https://www.clinicalkey.com/#!/content/book/3-s2.0-B9781455775668006050